CLINICAL TRIAL: NCT02345252
Title: A Phase 3b, Randomized, Double-Blind Switch Study to Evaluate the Safety and Efficacy of Emtricitabine/Rilpivirine/Tenofovir Alafenamide (FTC/RPV/TAF) Fixed Dose Combination (FDC) in HIV-1 Positive Subjects Who Are Virologically Suppressed on Emtricitabine/Rilpivirine/Tenofovir Disoproxil Fumarate (FTC/RPV/TDF)
Brief Title: Switch Study to Evaluate the Safety and Efficacy of Emtricitabine/Rilpivirine/Tenofovir Alafenamide (FTC/RPV/TAF) Fixed Dose Combination (FDC) in HIV-1 Positive Adults Who Are Virologically Suppressed on Emtricitabine/Rilpivirine/Tenofovir Disoproxil Fumarate (FTC/RPV/TDF)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GS-US-366-1216; 2014-004545-27 (EudraCT Number)
Record Dates: First submitted 2015-01-19; First posted 2015-01-26 (Estimated); Results first posted 2017-12-08 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: HIV-1 Infection
Keywords: HIV
MeSH Terms: interventions — Emtricitabine, Rilpivirine, Tenofovir Drug Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- FTC/RPV/TAF (Experimental): FTC/RPV/TAF plus FTC/RPV/TDF placebo for at least 96 weeks.
  Interventions: Drug: FTC/RPV/TAF; Drug: FTC/RPV/TDF Placebo
- FTC/RPV/TDF (Active Comparator): FTC/RPV/TDF plus FTC/RPV/TAF placebo for at least 96 weeks.
  Interventions: Drug: FTC/RPV/TDF; Drug: FTC/RPV/TAF Placebo
- Open Label Extension Phase (Experimental): After the Week 96 visit is completed, participants will be given the option to receive open label FTC/RPV/TAF for up to an additional 48 weeks. In countries where FTC/RPV/TAF is not yet commercially available, participants will be given the option to receive open-label FTC/RPV/TAF, and attend visits every 12 weeks until FTC/RPV/TAF becomes commercially available, or until Gilead Sciences elects to discontinue the study, whichever occurs first.
  Interventions: Drug: FTC/RPV/TAF

INTERVENTIONS:
Drug: FTC/RPV/TAF — 200/25/25 mg FDC tablets administered orally once daily
  Other Names: Odefsey®
  Arms: FTC/RPV/TAF; Open Label Extension Phase
Drug: FTC/RPV/TDF Placebo — Tablets administered orally once daily
  Arms: FTC/RPV/TAF
Drug: FTC/RPV/TDF — 200/25/300 mg FDC tablets administered orally once daily
  Other Names: Complera®; Eviplera®
  Arms: FTC/RPV/TDF
Drug: FTC/RPV/TAF Placebo — Tablets administered orally once daily
  Arms: FTC/RPV/TDF

SUMMARY:
The primary objective of this study is to evaluate the noninferiority of switching to emtricitabine/rilpivirine /tenofovir alafenamide (FTC/RPV/TAF) fixed-dose combination (FDC) as compared to continuing FTC/RPV/tenofovir disoproxil fumarate (TDF) FDC (FTC/RPV/TDF) in virologically suppressed HIV-1 infected participants.

ELIGIBILITY:
Key Inclusion Criteria:

* The ability to understand and sign a written informed consent form, which must be obtained prior to initiation of study procedures
* Currently receiving FTC/RPV/TDF FDC for ≥ 6 consecutive months preceding the screening visit
* Documented plasma HIV-1 RNA levels < 50 copies/mL (or undetectable HIV-1 RNA level according to the local assay being used if the limit of detection is > 50 copies/mL) for ≥ 6 months preceding the screening visit. After reaching HIV-1 RNA < 50 copies/mL, single values of HIV-1 RNA ≥ 50 copies/mL followed by resuppression, are allowed
* Have no documented resistance to any of the study agents at any time in the past
* HIV-1 RNA < 50 copies/mL at the screening visit
* Hepatic transaminases (AST and ALT) ≤ 5 × upper limit of normal (ULN)
* Total bilirubin ≤ 1.5 mg/dL (≤ 26 μmol/L), or normal direct bilirubin
* Adequate hematologic function (absolute neutrophil count ≥ 1,000/mm^3 (1.00 GI/L); platelets ≥ 50,000/mm^3 (50 GI/L); hemoglobin ≥ 8.5 g/dL (85 g/L))
* Serum amylase ≤ 5 × ULN (individuals with serum amylase > 5 × ULN will remain eligible if serum lipase is ≤ 5 × ULN)
* Normal ECG (or if abnormal, determined by the Investigator to be not clinically significant)
* Adequate renal function: Estimated glomerular filtration rate ≥ 50 mL/min (1.17 mL/sec) according to the Cockcroft-Gault formula

Key Exclusion Criteria:

* Hepatitis B surface antigen (HBsAg) positive
* Hepatitis C antibody positive with detectable hepatitis C virus (HCV) RNA (individuals who have HCV antibody but no detectable HCV RNA are eligible to enroll)
* Individuals experiencing or with a medical history of decompensated cirrhosis (e.g., ascites, encephalopathy, etc.)
* Females who are breastfeeding
* Positive serum pregnancy test
* Current alcohol or substance use judged by the Investigator to potentially interfere with individual's study compliance
* A history of malignancy within the past 5 years (prior to screening) or ongoing malignancy other than cutaneous Kaposi's sarcoma (KS), basal cell carcinoma, or resected, non-invasive cutaneous squamous carcinoma. Individuals with cutaneous KS are eligible, but must not have received any systemic therapy for KS within 30 days of Baseline/Day 1 and must not be anticipated to require systemic therapy during the study
* Active, serious infections (other than HIV-1 infection) requiring parenteral antibiotic or antifungal therapy within 30 days prior to Baseline/Day 1
* Any other clinical condition or prior therapy that, in the opinion of the Investigator, would make the individual unsuitable for the study or unable to comply with dosing requirements
* Participation in any other clinical trial (including observational trials) without prior approval from the sponsor is prohibited while participating in this trial
* Individuals receiving ongoing therapy with any of the disallowed medications listed in the protocol, including drugs not to be used with FTC, RPV and/or TAF; or individuals with any known allergies to the excipients of FTC/RPV/TAF

Note: Other Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 632 (Actual)
Dates: Start 2015-01-26 (Actual); Primary Completion 2016-06-22 (Actual); Study Completion 2019-01-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (117):
- United States (75):
  - The University of Alabama at Birmingham (UAB), Birmingham, Alabama
  - Spectrum Medical Group, Phoenix, Arizona
  - AHF Research Center, Beverly Hills, California
  - Pacific Oaks Medical Group, Beverly Hills, California
  - Long Beach Education and Research Consultants, Long Beach, California
  - Kaiser Permanente, Los Angeles, California
  - Southern California Men's Medical Group, Los Angeles, California
  - Tarrant County ID Associates, Los Angeles, California
  - Alameda County Medical Center, Oakland, California
  - Desert Medical Group Inc., dba Desert Oasis Healthcare Medical Group, Palm Springs, California
  - Kaiser Permanente, Sacramento, California
  - University of California-UC Davis, Sacramento, California
  - La Playa Medical Group and Clinical Research, San Diego, California
  - Kaiser Permanente, San Francisco, California
  - Optimus Medical, San Francisco, California
  - Kaiser Permanente, San Leandro, California
  - Los Angeles BioMedical Institute at Harbor-UCLA Medical Center, Torrance, California
  - University of Colorado, Aurora, Colorado
  - Apex Research Institute, Denver, Colorado
  - Yale University School of Medicine, New Haven, Connecticut
  - World Health Clinicians' CIRCLE CARE Center, Norwalk, Connecticut
  - Capital Medical Associates, P.C., Washington D.C., District of Columbia
  - Dupont Circle Physicians Group, Washington D.C., District of Columbia
  - Medical Faculty Associates, Washington D.C., District of Columbia
  - Whitman Walker Clinic, Washington D.C., District of Columbia
  - Gary Richmond, MD, PA, Inc., Fort Lauderdale, Florida
  - Therafirst Medical Centers, Fort Lauderdale, Florida
  - Midway Immunology & Research Center, LLC, Ft. Pierce, Florida
  - AIDS Healthcare Foundation, Miami, Florida
  - AIDS Healthcare Foundation, Miami Beach, Florida
  - Orlando Immunology Center, Orlando, Florida
  - Infectious Diseases Associates of NW Florida, P.A., Pensacola, Florida
  - Hillsborough County Health Dept., Tampa, Florida
  - Infectious Disease Research Institute Inc., Tampa, Florida
  - St. Joseph's Comprehensive Research Institute, Tampa, Florida
  - AIDS Research & Treatment Center of the Treasure Coast, Vero Beach, Florida
  - Triple O Research Institute, P.A., West Palm Beach, Florida
  - Rowan Tree Medical PA, Wilton Manors, Florida
  - AIDS Research Consortium of Atlanta, Atlanta, Georgia
  - Atlanta ID Group, Atlanta, Georgia
  - Infectious Disease Specialists of Atlanta, Decatur, Georgia
  - Chatham County Health Department, Savannah, Georgia
  - Indiana University Medical Center, Indianapolis, Indiana
  - Brigham and Women's, Boston, Massachusetts
  - Community Research Initiative, Boston, Massachusetts
  - MetroWest Medical Center, Framingham, Massachusetts
  - Baystate Infectious Diseases Clinical Research, Springfield, Massachusetts
  - The Research Institute, Springfield, Massachusetts
  - Be Well Medical Center, Berkley, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Southampton Healthcare, Inc., St Louis, Missouri
  - Jersey Shore Medical Center, Neptune City, New Jersey
  - Saint Michael's Medical Center, Newark, New Jersey
  - South Jersey Infectious Disease, Somers Point, New Jersey
  - Southwest CARE Center, Santa Fe, New Mexico
  - Upstate Infectious Diseases Associates, Albany, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Carolinas Medical Center--Myers Park Infectious Disease Clinic, Charlotte, North Carolina
  - Rosedale Infectious Diseases, Huntersville, North Carolina
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Central Texas Clinical Research, Austin, Texas
  - North Texas Infectious Diseases Consultants, Dallas, Texas
  - Trinity Health and Wellness Center/AIDS Arms, Inc., Dallas, Texas
  - AIDS Arms, Inc./Trinity Health & Wellness Center, Fort Worth, Texas
  - Gordon E. Crofoot, MD, PA, Houston, Texas
  - Research Access Network, Houston, Texas
  - DCOL Center for Clinical Research, Longview, Texas
  - Clinical Alliance for Research & Education - Infectious Diseases, LLC (CARE-ID), Annandale, Virginia
  - Peter Shalit, MD, Seattle, Washington
  - Premier Clinical Research, Spokane, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Belgium (3):
  - CHU Saint-Pierre University Hospital, Brussels
  - Cliniques Universitaires UCL Saint-Luc, Brussels
  - University Hospital Gent, Ghent
- Canada (7):
  - University of Alberta, Edmonton, Alberta
  - Spectrum Health, Vancouver, British Columbia
  - Maple Leaf Research, Toronto, Ontario
  - University Health Network, Toronto, Ontario
  - Clinique medicale l'Actuel, Montreal, Quebec
  - Clinique OPUS, Montreal, Quebec
  - McGill University Health Centre, Montreal, Quebec
- Hôpital Gui de Chauliac - Service Maladies Infectieuses et Tropicales, Montpellier, France
- Germany (10):
  - Zentrum für Infektiologie Berlin Prenzlauer Berg GmbH (zibp), Berlin
  - University of Bonn, Bonn
  - Universitat zu Koln, Cologne
  - Center for HIV and Hepatogastroenterology, Düsseldorf
  - Universitätsklinikum Essen, Essen
  - Infektiologikum, Frankfurt
  - Asklepios Klinik, Hamburg
  - ICH Study Center Hamburg, Hamburg
  - Universitatsklinikum Hamburg-Eppendorf, Hamburg
  - MUC Research GmbH, München
- Italy (2):
  - Azienda Ospedaliera Papa Giovanni XXIII, Bergamo
  - Fondazione IRCCS San Raffaele del Monte Tabor, Milan
- Erasmus MC, Rotterdam, Netherlands
- Puerto Rico (2):
  - Clinical Research Puerto Rico Inc, San Juan
  - Hope Clinical Research, San Juan
- Spain (7):
  - Hospital General Universitario de Alicante, Alicante
  - Hospital Germans Trias i Pujol, Badalona
  - Hospital del Mar, Barcelona
  - Hospital Universitary de Bellvitge, Barcelona
  - Hospital Clínico Universitario San Carlos, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
- Karolinska Institutet, Stockholm, Sweden
- Switzerland (2):
  - University Hospital Basel, Basel
  - Geneva University Hospital, Geneva
- United Kingdom (6):
  - NHS Greater Glasgow, Glasgow
  - Barts & The London NHS Trust, London
  - Chelsea & Westminster Hospital, London
  - Mortimer Market Centre, London
  - The Royal Free Hampstead NHS Trust, London
  - The Hathersage Integrated Contraception, Sexual Health and HIV Service, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Qualified external researchers may request IPD for this study after study completion. For more information, please visit our website at http://www.gilead.com/research/disclosure-and-transparency.
Supporting Information: Study Protocol, SAP
Time Frame: 18 months after study completion
Access Criteria: A secured external environment with username, password, and RSA code.
URL: http://www.gilead.com/research/disclosure-and-transparency

REFERENCES:
- [Result] Hagins D, Orkin C, Daar ES, Mills A, Brinson C, DeJesus E, Post FA, Morales-Ramirez J, Thompson M, Osiyemi O, Rashbaum B, Stellbrink HJ, Martorell C, Liu H, Liu YP, Porter D, Collins SE, SenGupta D, Das M. Switching to coformulated rilpivirine (RPV), emtricitabine (FTC) and tenofovir alafenamide from either RPV, FTC and tenofovir disoproxil fumarate (TDF) or efavirenz, FTC and TDF: 96-week results from two randomized clinical trials. HIV Med. 2018 Nov;19(10):724-733. doi: 10.1111/hiv.12664. Epub 2018 Aug 12. PMID 30101539
- [Result] Mills A, Brinson C, Martorell C, Crofoot G, Daar E, Osiyemi O, et al. Switching to RPV/FTC/TAF from RPV/FTC/TDF or EFV/FTC/TDF: Week 96 Results. Conference on Retroviruses and Opportunistic Infections,Boston. March 4-7, 2018, Abstract 504.
- [Result] Arribas JR, Rockstroh J, Post, Yazdanpanah Y, Cavassini, DeJesus E, et al. Bone and renal safety of switching to rilpivirine/emtricitabine/tenofovir alafenamide (RPV/FTC/TAF) from single-tablet regimens (STRs) containing efavirenz/emtricitabine/tenofovir disoproxil fumarate (EFV/FTC/TDF) or rilpivirine/emtricitabine/tenofovir disoproxil fumarate (RPV/FTC/TDF): Week48 subgroup analysis in patients at risk of or with comorbidities. Abstract accepted for presentation atthe 16th European AIDS Conference, 2017 25-27 October Milan, Italy.
- [Result] Porter DP, Kulkarni R, Cao H, SenGupta D, White KL. No Emergent Resistance in HIV-1 Virologically-Suppressed Subjects Who Switched to RPV/FTC/TAF [Poster1381]. ID Week™ (Infectious Diseases Society of America) 2017 4-8 October; San Diego, CA.
- [Result] Wohl D, Kulkarni R, Garner W, White KL, Porter DL. Viral Blips Were Infrequent in HIV1-Infected Virologically-Suppressed Adults Treated with Tenofovir Alafenamide or Tenofovir DF Rilpivirine-Containing Regimens [Poster1384]. ID Week™ (Infectious Diseases Society of America) 2017 4-8 October; San Diego, CA.
- [Result] DeJesus E, Ramgopal M, Crofoot G, Ruane P, LaMarca A, Molina J-M, et al. Efficacy and Safety of Switching to RPV/FTC/TAF in Older Adults. 8th International Workshopon HIV and Aging 2017 2-3 October, New York, New York.
- [Result] Molina JM, DeJesus E, Rijnders B, Post FAV, B., Stoeckle M, Thalme A, et al. Efficacy and Odefsey® StudyGS-US-366-1216Final Synoptic Clinical Study Report Final CONFIDENTIAL Page4 30July2019 Safety of Switching From RPV/FTC/TDF or EFV/FTC/TDF to RPV/FTC/TAF in Black Adults [Presentation MOPEB0291]. 9th IAS Conference on HIV Science 2017 23-26 July Paris, France.
- [Result] Rockstroh J, Orkin C, Yazdanpanah Y, Di Perri GDS, P. E., Arribas JR, Brinkman K, et al. Switching From TDF to TAF Improves Bone and Renal Safety Independent of Age, Sex, Race, or 3rd Agent: Results From Pooled Analysis (N=3816) of Virologically Suppressed HIV-1 Infected Adults [Presentation MOPEB0289]. 9th IAS Conference on HIV Science;2017 23-26July Paris, France.
- [Result] Orkin C, DeJesus E, Ramgopal M, Crofoot G, Ruane P, LaMarca A, Mills A, Vandercam B, de Wet J, Rockstroh J, Lazzarin A, Rijnders B, Podzamczer D, Thalme A, Stoeckle M, Porter D, Liu HC, Cheng A, Quirk E, SenGupta D, Cao H. Switching from tenofovir disoproxil fumarate to tenofovir alafenamide coformulated with rilpivirine and emtricitabine in virally suppressed adults with HIV-1 infection: a randomised, double-blind, multicentre, phase 3b, non-inferiority study. Lancet HIV. 2017 May;4(5):e195-e204. doi: 10.1016/S2352-3018(17)30031-0. Epub 2017 Mar 2. PMID 28259777
- [Result] Majeed SR, Shao Y, Garner W, Scott J, Pérez-Ruixo C, SenGupta D, et al. Evaluation of RPV/FTC/TAF Exposure-Efficacy and Exposure-Safety Relationships [Poster427]. Conference on Retroviruses and Opportunistic Infections (CROI) 2017 13-16 February; Seattle, WA.
- [Result] Hagins D, Mills A, Martorell C, Walmsley S, Gallant J, Tebas P, et al. Efficacy and Safety of Switching toRPV/FTC/TAF in Women [Abstract12]. 7th International Workshop on HIV & Women; 2017 11-12 February; Seattle, Washington.
- [Result] Orkin C, DeJesus E, Ramgopal M, Crofoot G, Ruane P, LaMarca A, et al. 48Week Results from two studies: Switching to RPV/FTC/TAF from EFV/FTC/TDF (Study1160) or RPV/FTC/TDF (Study1216) [Presentation]. HIV Glasgow; 2016 23-26 October; Glasgow, United Kingdom.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in Europe and North America. The first participant was screened on 26 January 2015. The last study visit occurred on 09 January 2019.
Pre-assignment Details: 690 participants were screened.
Groups:
- FTC/RPV/TAF: Double-Blind Phase: Emtricitabine/rilpivirine/tenofovir alafenamide (FTC/RPV/TAF) (200/25/25 mg) fixed-dose combination (FDC) tablet + emtricitabine/rilpivirine/tenofovir disoproxil fumarate (FTC/RPV/TDF) placebo tablet orally once daily for up to 96 weeks.
  Open-Label Extension Phase: After the Week 96 visit, participants were given the option to receive open label FTC/RPV/TAF FDC for up to an additional 48 weeks. In countries where FTC/RPV/TAF FDC was not yet commercially available, participants were given the option to receive open-label FTC/RPV/TAF FDC orally once daily attend visits every 12 weeks until FTC/RPV/TAF FDC became commercially available, or until Gilead elected to discontinue the study, whichever occurred first.
- FTC/RPV/TDF: Double-Blind Phase: FTC/RPV/TDF (200/25/300 mg) FDC tablet + FTC/RPV/TAF placebo tablet orally once daily for up to 96 weeks.
  Open-Label Extension Phase: After the Week 96 visit, participants were given the option to receive open label FTC/RPV/TAF FDC for up to an additional 48 weeks. In countries where FTC/RPV/TAF FDC was not yet commercially available, participants were given the option to receive open-label FTC/RPV/TAF FDC orally once daily and attend visits every 12 weeks until FTC/RPV/TAF FDC became commercially available, or until Gilead elected to discontinue the study, whichever occurred first.
Period: Double-Blind Phase
Arm/Group | FTC/RPV/TAF | FTC/RPV/TDF
Started | 316 | 316
Completed | 276 | 267
Not Completed | 40 | 49
Not completed — Adverse Event | 2 | 3
Not completed — Death | 1 | 2
Not completed — Lack of Efficacy | 1 | 0
Not completed — Investigator's Discretion | 4 | 6
Not completed — Non-Compliance with Study Drug | 1 | 2
Not completed — Protocol Violation | 2 | 1
Not completed — Withdrew Consent | 21 | 23
Not completed — Lost to Follow-up | 8 | 10
Not completed — Randomized but Never Treated | 0 | 2
Period: Open-Label Extension Phase
Arm/Group | FTC/RPV/TAF | FTC/RPV/TDF
Started | 19 (257 participants completed the Double-Blind Phase, but did not enter Open-Label Extension Phase.) | 17 (250 participants completed the Double-Blind Phase, but did not enter Open-Label Extension Phase.)
Completed | 19 | 17
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set included participants who were randomized and received at least 1 dose of study drug.
Groups:
- FTC/RPV/TAF: FTC/RPV/TAF (200/25/25 mg) FDC tablet + FTC/RPV/TDF placebo tablet orally once daily for up to 96 weeks.
- FTC/RPV/TDF: FTC/RPV/TDF (200/25/300 mg) FDC tablet + FTC/RPV/TAF placebo tablet orally once daily for up to 96 weeks.
- Total: Total of all reporting groups
Arm/Group | FTC/RPV/TAF | FTC/RPV/TDF | Total
Number analyzed (Participants) | 316 | 314 | 630
Age, Continuous [Mean (Standard Deviation); unit: years] | 45 (10.4) | 44 (10.2) | 45 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 25 | 66
  Male | 275 | 289 | 564
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 2 | 3
  Asian | 7 | 17 | 24
  Black | 65 | 54 | 119
  Native Hawaiian or Pacific Islander | 0 | 1 | 1
  White | 238 | 235 | 473
  Other | 5 | 5 | 10
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 40 | 53 | 93
  Not Hispanic or Latino | 275 | 261 | 536
  Not Permitted | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 24 | 11 | 35
  Netherlands | 3 | 4 | 7
  Sweden | 2 | 2 | 4
  Belgium | 5 | 4 | 9
  United States | 222 | 226 | 448
  Italy | 3 | 8 | 11
  United Kingdom | 10 | 9 | 19
  France | 1 | 1 | 2
  Switzerland | 4 | 4 | 8
  Germany | 27 | 30 | 57
  Spain | 15 | 15 | 30
HIV-1 RNA Category [Count of Participants; unit: Participants]
  < 50 copies/mL | 307 | 312 | 619
  ≥ 50 copies/mL | 9 | 2 | 11
CD4 Cell Count [Mean (Standard Deviation); unit: cells/μL] | 711 (278.9) | 707 (264.7) | 709 (271.7)
CD4 Cell Count Category [Count of Participants; unit: Participants]
  ≥ 50 to < 200 cells/µL | 5 | 1 | 6
  ≥ 200 to < 350 cells/µL | 10 | 16 | 26
  ≥ 350 to < 500 cells/µL | 52 | 50 | 102
  ≥ 500 cells/ µL | 249 | 247 | 496

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With HIV-1 RNA < 50 Copies/mL at Week 48 as Defined by the US FDA-Defined Snapshot Algorithm
Description: The percentage of participants achieving HIV-1 RNA < 50 copies/mL at Week 48 was analyzed using the US FDA-defined snapshot algorithm, which defines a patient's virologic response status using only the viral load at the predefined time point within an allowed window of time, along with study drug discontinuation status.
Time Frame: Week 48
Population: The Full Analysis Set included participants who were randomized and received at least 1 dose of study drug and were on FTC/RPV/TDF prior to the screening visit.
Measure: Number; unit: percentage of participants
Arm/Group | FTC/RPV/TAF | FTC/RPV/TDF
Number analyzed (Participants) | 316 | 313
percentage of participants | 93.7 | 93.9
Statistical Analysis 1: Comparison: FTC/RPV/TAF vs FTC/RPV/TDF; The null hypothesis was that the percentage of participants with HIV-1 RNA < 50 copies/mL at Week 48 in the FTC/RPV/TAF group was at least 8% lower than the rate in the FTC/RPV/TDF group; the alternative hypothesis was that the percentage of participants with HIV-1 RNA < 50 copies/mL in the FTC/RPV/TAF group was less than 8% lower than that in the FTC/RPV/TDF group; Test type: Non-Inferiority — A sample size of 275 HIV-1 infected participants per treatment group would provide 85% power to detect a noninferiority margin of 8% in the Week 48 response rate difference between the FTC/RPV/TAF group and FTC/RPV/TDF group. For sample size and power computation, it is assumed that both treatment groups will have a response rate of 89% (based on Gilead Study GS-US-292-0109), that a noninferiority margin is 8%, and that the significance level of the test is at a one-sided alpha level of 0.025; Difference in Percentages = -0.3, 95.001% CI 2-sided [-4.2 to 3.7] — The difference in percentages and its 95.001% confidence interval (CI) were calculated based on an unconditional exact method using 2 inverted 1-sided tests
Statistical Analysis 2: Comparison: FTC/RPV/TAF vs FTC/RPV/TDF; Test type: Superiority; p = 1.00, Fisher Exact

2. Secondary Outcome: Percentage of Participants With HIV-1 RNA ≥ 50 Copies/mL at Week 48 as Defined by the US FDA-Defined Snapshot Algorithm
Description: The percentage of participants with HIV-1 RNA ≥ 50 copies/mL at Week 48 was analyzed using the snapshot algorithm, which defines a patient's virologic response status using only the viral load at the predefined time point within an allowed window of time, along with study drug discontinuation status.
Time Frame: Week 48
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | FTC/RPV/TAF | FTC/RPV/TDF
Number analyzed (Participants) | 316 | 313
percentage of participants | 0.6 | 0

3. Secondary Outcome: Percentage of Participants With HIV-1 RNA ≥ 50 Copies/mL at Week 96 as Defined by the US FDA-Defined Snapshot Algorithm
Description: The percentage of participants with HIV-1 RNA ≥ 50 copies/mL at Week 96 was analyzed using the snapshot algorithm, which defines a patient's virologic response status using only the viral load at the predefined time point within an allowed window of time, along with study drug discontinuation status.
Time Frame: Week 96
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | FTC/RPV/TAF | FTC/RPV/TDF
Number analyzed (Participants) | 316 | 313
percentage of participants | 0.6 | 1.0

4. Secondary Outcome: Percentage of Participants With HIV-1 RNA < 50 Copies/mL at Week 96 as Defined by the US FDA-Defined Snapshot Algorithm
Description: The percentage of participants with HIV-1 RNA < 50 copies/mL at Week 96 was analyzed using the snapshot algorithm, which defines a patient's virologic response status using only the viral load at the predefined time point within an allowed window of time, along with study drug discontinuation status.
Time Frame: Week 96
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | FTC/RPV/TAF | FTC/RPV/TDF
Number analyzed (Participants) | 316 | 313
percentage of participants | 89.2 | 88.5

5. Secondary Outcome: Change From Baseline in CD4+ Cell Count at Week 48
Time Frame: Baseline; Week 48
Population: Participants in the Full Analysis Set with on-treatment data were analyzed.
Measure: Mean (Standard Deviation); unit: cells/µL
Arm/Group | FTC/RPV/TAF | FTC/RPV/TDF
Number analyzed (Participants) | 296 | 293
cells/µL | 9 (159.7) | -1 (152.7)

6. Secondary Outcome: Change From Baseline in CD4+ Cell Count at Week 96
Time Frame: Baseline; Week 96
Population: Participants in the Full Analysis Set with on-treatment data were analyzed.
Measure: Mean (Standard Deviation); unit: cells/µL
Arm/Group | FTC/RPV/TAF | FTC/RPV/TDF
Number analyzed (Participants) | 283 | 277
cells/µL | 12 (180.6) | 16 (171.9)

7. Secondary Outcome: Percent Change From Baseline in Hip Bone Mineral Density (BMD) at Week 48
Description: Hip BMD was assessed by dual energy x-ray absorptiometry (DXA) scan.
Time Frame: Baseline; Week 48
Population: Participants in the Hip DXA Analysis Set (all randomized participants who received at least 1 dose of study drug, and had nonmissing baseline hip BMD value) with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | FTC/RPV/TAF | FTC/RPV/TDF
Number analyzed (Participants) | 168 | 165
percentage change | 1.040 (1.9404) | -0.245 (2.0805)

8. Secondary Outcome: Percent Change From Baseline in Hip BMD at Week 96
Description: Hip BMD was assessed by DXA scan.
Time Frame: Baseline; Week 96
Population: Participants in the Hip DXA Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | FTC/RPV/TAF | FTC/RPV/TDF
Number analyzed (Participants) | 160 | 156
percentage change | 1.623 (2.4575) | -0.613 (2.7411)

9. Secondary Outcome: Percent Change From Baseline in Spine BMD at Week 48
Description: Spine BMD was assessed by DXA scan.
Time Frame: Baseline; Week 48
Population: Participants in the spine DXA Analysis Set (all randomized participants who received at least 1 dose of study drug, and had nonmissing baseline hip BMD value) with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | FTC/RPV/TAF | FTC/RPV/TDF
Number analyzed (Participants) | 172 | 168
percentage change | 1.613 (3.4346) | 0.075 (2.9605)

10. Secondary Outcome: Percent Change From Baseline in Spine BMD at Week 96
Description: Spine BMD was assessed by DXA scan.
Time Frame: Baseline; Week 96
Population: Participants in the Spine DXA Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | FTC/RPV/TAF | FTC/RPV/TDF
Number analyzed (Participants) | 162 | 158
percentage change | 2.039 (3.5098) | -0.250 (3.5903)

ADVERSE EVENTS:
Time Frame: First dose date to last dose date (maximum duration: 173.1 weeks) plus 30 days
Description: The Safety Analysis Set included participants who were randomized and received at least 1 dose of study drug.
Groups:
- FTC/RPV/TAF (Double-Blind Phase): Adverse events reported occurred during the Double-Blind Phase in participants from the FTC/RPV/TAF group, who received FTC/RPV/TAF (200/25/25 mg) FDC tablet plus FTC/RPV/TDF placebo tablet administered orally once daily.
- FTC/RPV/TDF (Double-Blind Phase): Adverse events reported occurred during the Double-Blind Phase in participants from the FTC/RPV/TDF group, who received FTC/RPV/TDF (200/25/300 mg) FDC tablet plus FTC/RPV/TAF placebo tablet administered orally once daily.
- Open-Label FTC/RPV/TAF From FTC/RPV/TAF: Adverse events reported occurred during the Open-Label Extension Phase in participants who enrolled into the Open-Label Extension Phase from the FTC/RPV/TAF group and received FTC/RPV/TAF (200/25/25 mg) FDC tablet once daily.
- Open-Label FTC/RPV/TAF From FTC/RPV/TDF: Adverse events reported occurred during the Open-Label Extension Phase in participants who enrolled into the Open-Label Extension Phase from the FTC/RPV/TDF group and received FTC/RPV/TAF (200/25/25 mg) FDC tablet once daily.
Arm/Group | FTC/RPV/TAF (Double-Blind Phase) | FTC/RPV/TDF (Double-Blind Phase) | Open-Label FTC/RPV/TAF From FTC/RPV/TAF | Open-Label FTC/RPV/TAF From FTC/RPV/TDF
All-Cause Mortality (participants affected / at risk) | 1/316 | 2/314 | 0/19 | 0/17
Serious Adverse Events (participants affected / at risk) | 36/316 | 29/314 | 1/19 | 0/17
Other Adverse Events (participants affected / at risk) | 249/316 | 234/314 | 14/19 | 11/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | FTC/RPV/TAF (Double-Blind Phase) (N=316) | FTC/RPV/TDF (Double-Blind Phase) (N=314) | Open-Label FTC/RPV/TAF From FTC/RPV/TAF (N=19) | Open-Label FTC/RPV/TAF From FTC/RPV/TDF (N=17)
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 0
Angina pectoris (Cardiac disorders) | 1 | 1 | 0 | 0
Angina unstable (Cardiac disorders) | 0 | 1 | 0 | 0
Coronary artery disease (Cardiac disorders) | 1 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastric ulcer perforation (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Chest pain (General disorders) | 1 | 0 | 0 | 0
Generalised oedema (General disorders) | 1 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 0 | 0
Bile duct stone (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 1 | 0 | 0
Abscess limb (Infections and infestations) | 1 | 0 | 0 | 0
Anal chlamydia infection (Infections and infestations) | 1 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 1 | 4 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 3 | 0 | 0 | 0
Cellulitis staphylococcal (Infections and infestations) | 1 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 2 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 0
Gastroenteritis cryptosporidial (Infections and infestations) | 1 | 0 | 0 | 0
Helicobacter infection (Infections and infestations) | 1 | 0 | 0 | 0
Hepatitis A (Infections and infestations) | 0 | 1 | 0 | 0
Myelitis (Infections and infestations) | 1 | 0 | 0 | 0
Osteomyelitis (Infections and infestations) | 2 | 0 | 0 | 0
Osteomyelitis acute (Infections and infestations) | 0 | 1 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 1 | 0 | 0
Proctitis gonococcal (Infections and infestations) | 1 | 0 | 0 | 0
Sepsis (Infections and infestations) | 1 | 1 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 1 | 0 | 0
Syphilis (Infections and infestations) | 1 | 0 | 0 | 0
Tooth abscess (Infections and infestations) | 0 | 1 | 0 | 0
Carbon monoxide poisoning (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Hyphaema (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Carotid artery aneurysm (Nervous system disorders) | 1 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 2 | 0 | 0 | 0
Cervicobrachial syndrome (Nervous system disorders) | 0 | 1 | 0 | 0
Paraplegia (Nervous system disorders) | 0 | 1 | 0 | 0
Completed suicide (Psychiatric disorders) | 0 | 1 | 0 | 0
Depression (Psychiatric disorders) | 1 | 1 | 0 | 0
Depression suicidal (Psychiatric disorders) | 1 | 0 | 0 | 0
Major depression (Psychiatric disorders) | 1 | 0 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 2 | 1 | 0 | 0
Suicide attempt (Psychiatric disorders) | 0 | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 1 | 0 | 0
Calculus urethral (Renal and urinary disorders) | 1 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0 | 0
Renal colic (Renal and urinary disorders) | 1 | 0 | 0 | 0
Priapism (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0 | 0
Pulmonary granuloma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Substance use (Social circumstances) | 1 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 2 | 0 | 0 | 0
Peripheral artery occlusion (Vascular disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | FTC/RPV/TAF (Double-Blind Phase) (N=316) | FTC/RPV/TDF (Double-Blind Phase) (N=314) | Open-Label FTC/RPV/TAF From FTC/RPV/TAF (N=19) | Open-Label FTC/RPV/TAF From FTC/RPV/TDF (N=17)
Lymphadenopathy (Blood and lymphatic system disorders) | 5 | 3 | 1 | 0
Hypothyroidism (Endocrine disorders) | 1 | 1 | 1 | 0
Blepharitis (Eye disorders) | 0 | 1 | 1 | 0
Conjunctivitis allergic (Eye disorders) | 0 | 0 | 2 | 0
Eye pain (Eye disorders) | 0 | 1 | 0 | 1
Meibomianitis (Eye disorders) | 0 | 0 | 1 | 0
Retinal detachment (Eye disorders) | 1 | 1 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 6 | 6 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 34 | 40 | 1 | 2
Flatulence (Gastrointestinal disorders) | 5 | 8 | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 2 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 20 | 11 | 0 | 0
Vomiting (Gastrointestinal disorders) | 17 | 10 | 0 | 0
Fatigue (General disorders) | 17 | 28 | 0 | 0
Influenza like illness (General disorders) | 2 | 3 | 1 | 0
Pyrexia (General disorders) | 7 | 13 | 0 | 3
Seasonal allergy (Immune system disorders) | 7 | 5 | 1 | 0
Anal chlamydia infection (Infections and infestations) | 3 | 9 | 1 | 0
Bronchitis (Infections and infestations) | 22 | 23 | 1 | 0
Chlamydial infection (Infections and infestations) | 10 | 8 | 1 | 0
Fungal skin infection (Infections and infestations) | 3 | 4 | 1 | 0
Gastroenteritis (Infections and infestations) | 10 | 11 | 1 | 0
Genital herpes (Infections and infestations) | 3 | 5 | 1 | 0
Influenza (Infections and infestations) | 19 | 18 | 0 | 0
Nasopharyngitis (Infections and infestations) | 49 | 46 | 0 | 3
Onychomycosis (Infections and infestations) | 4 | 6 | 1 | 0
Oral herpes (Infections and infestations) | 6 | 3 | 2 | 0
Papilloma viral infection (Infections and infestations) | 2 | 2 | 1 | 0
Pharyngitis (Infections and infestations) | 14 | 13 | 1 | 0
Pneumonia (Infections and infestations) | 1 | 6 | 1 | 0
Respiratory tract infection (Infections and infestations) | 3 | 2 | 0 | 1
Rhinitis (Infections and infestations) | 5 | 2 | 0 | 1
Sinusitis (Infections and infestations) | 20 | 23 | 0 | 0
Syphilis (Infections and infestations) | 16 | 23 | 0 | 0
Tooth infection (Infections and infestations) | 5 | 6 | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 47 | 46 | 1 | 1
Contusion (Injury, poisoning and procedural complications) | 10 | 5 | 1 | 0
Post-traumatic pain (Injury, poisoning and procedural complications) | 1 | 3 | 0 | 1
Weight decreased (Investigations) | 3 | 3 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 24 | 32 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 28 | 34 | 2 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 4 | 4 | 0 | 1
Muscle contracture (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 10 | 9 | 0 | 2
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 11 | 4 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 25 | 16 | 1 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 2 | 0
Dizziness (Nervous system disorders) | 11 | 11 | 0 | 1
Facial paralysis (Nervous system disorders) | 0 | 3 | 0 | 1
Headache (Nervous system disorders) | 25 | 24 | 0 | 2
Paraesthesia (Nervous system disorders) | 8 | 7 | 1 | 0
Sciatica (Nervous system disorders) | 4 | 1 | 1 | 0
Syncope (Nervous system disorders) | 2 | 2 | 1 | 0
Anxiety (Psychiatric disorders) | 17 | 13 | 0 | 1
Depressed mood (Psychiatric disorders) | 1 | 2 | 0 | 1
Depression (Psychiatric disorders) | 20 | 13 | 0 | 0
Insomnia (Psychiatric disorders) | 11 | 18 | 0 | 1
Sleep sex (Psychiatric disorders) | 0 | 0 | 0 | 1
Dysuria (Renal and urinary disorders) | 5 | 5 | 1 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 9 | 1 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 6 | 4 | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 22 | 24 | 2 | 3
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 8 | 3 | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 6 | 4 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 2 | 1 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 1 | 2 | 1 | 0
Skin fissures (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0
Hypertension (Vascular disorders) | 22 | 9 | 0 | 0
Varicose vein (Vascular disorders) | 2 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years